CLINICAL TRIAL: NCT02966730
Title: Protocol 20060 (PCYC): A Multicenter, Open-Label Pilot Study of Follicular Lymphoma Ibrutinib Consolidation for FDG-PET Positivity After Frontline Chemoimmunotherapy (FLIPP)
Brief Title: Ibrutinib for Patients With Follicular Lymphoma Without Complete Response to Initial Chemoimmunotherapy
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Fox Chase Cancer Center (Other); Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-396
Record Dates: First submitted 2016-11-14; First posted 2016-11-17 (Estimated); Last update posted 2025-05-13 (Actual); Status verified 2019-06

CONDITIONS: Follicular Lymphoma; Follicular Lymphoma, Grade 1; Follicular Lymphoma, Grade 2; Follicular Lymphoma Grade IIIa
Keywords: follicular lymphoma; Ibrutinib; FLIPP; 16-396
MeSH Terms: conditions — Lymphoma, Follicular | interventions — ibrutinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (1):
- Follicular Lymphoma (Experimental): Participants will be receive Ibrutinib as an oral capsule preparation once daily for a period of 2 years. The dose will be 560mg daily. Toxicities will be recorded and graded. Response to treatment will be determined by FDG-PET imaging every 6 months, or as clinically indicated, in conjunction with clinical assessment by a physician, including physical examination, every 4 weeks from day 1 (baseline) for the first 3 months and then every 3 months until the end of treatment at 2 years.
  Interventions: Drug: Ibrutinib

INTERVENTIONS:
Drug: Ibrutinib — Ibrutinib will be administered orally, on a once daily continuous dosing schedule and in an outpatient setting. Treatment will continue for 2 years and there will be no planned treatment breaks. The dose of Ibrutinib will be initiated at 560mg per day, which will remain constant throughout the study period, unless otherwise specified.

SUMMARY:
The purpose of this study is to find out how successful ibrutinib is at putting follicular lymphoma into full remission. In this study, remission will be determined by achieving a normal PET scan after treatment. A PET scan is an imaging test that looks for active lymphoma. People who don't have a complete remission on PET after their first treatment are at high risk for having their lymphoma return. This study will investigate if ibrutinib will help participants achieve a complete remission without giving additional chemotherapy. The study will also investigate any possible side effects of the study drug ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Follicular lymphoma with histology documented by the participating institution (grades 1, 2 or 3a).

  °For subjects with presumptive evidence of transformation based on clinical assessment of factors such as, but not limited to, increasing lactate dehydrogenase (LDH), rapidly worsening disease, or frequent B-symptoms, a pre-treatment biopsy is required to rule out large cell transformation
* Completion of a full course of first line immunochemotherapy including rituximab OR completion of 4 cycles of first line immunochemotherapy including rituximab if intolerant (e.g. which include, but are not limited to, R-CHOP, R-CVP, Bendamustine-R).
* Patients must have achieved PR to primary treatment and not be refractory to prior treatment.
* Residual FDG-PET activity defined as Deauville 4 or 5 on a PET-CT within 3 and 8 weeks post the last dose of front line therapy.
* Treatment must begin within 90 days of the last dose of immunochemotherapy.
* Men and women ≥ 18 years of age.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2.
* ≥ 1 measurable disease site on computed tomography (CT) scan or positron emission tomography (PET) (1.5 cm in longest dimension). (In select cases, for example extremity lesions, an MRI may be substituted.)
* Life expectancy of > 3 months, in the opinion of the investigator.
* Female subjects who are of non-reproductive potential (i.e. post-menopausal by history - no menses for ≥ 2 years; OR history of hysterectomy; OR history of bilateral tubal ligation; OR history of bilateral oophorectomy). Female subjects of childbearing potential must have a negative serum pregnancy test upon study entry.
* Male and female subjects who agree to use highly effective methods of birth control (e.g., implants, injectables, combined oral contraceptives, some intrauterine devices [IUDs], sexual abstinence, or sterilized partner) and a barrier method (e.g. condoms, vaginal ring, sponge, etc) during the period of therapy and for 30 days (females) and 90 days (males) after the last dose of study drug.

Exclusion Criteria:

* Medically apparent central nervous system lymphoma or leptomeningeal disease.
* History of any other active malignancies.
* History of any prior cancer curatively treated within the last two years except:

  * Any non-melanoma skin cancer
  * Any cancer excised, not treated with chemotherapy and with less than a 30% chance of recurrence within the next 2 years from registration
* History of any organ transplantation.
* History of stroke or intracranial hemorrhage within 6 months prior to enrollment.
* More than one prior line of any systemic chemoimmunotherapy for follicular lymphoma.
* Chemotherapy ≤ 21 days prior to first administration of study treatment and/or monoclonal antibody ≥ 3 weeks prior to first administration of study treatment.
* Prior exposure to radio- or toxin-immunoconjugates.
* Concurrent use of warfarin or other vitamin K antagonists.
* Concurrent use of a strong cytochrome P450 (CYP)3A4/5 inhibitor.
* Concurrent systemic immunosuppressant therapy (e.g., cyclosporine A, tacrolimus, etc., or chronic administration of > 20 mg/day of prednisone) within 28 days of the first dose of study drug.
* Vaccinated with live, attenuated vaccines within 4 weeks of first dose of study drug.
* Significant screening electrocardiogram (ECG) abnormalities including left bundle branch block, 2nd degree atrioventricular (AV) block type II, 3rd degree block, or corrected QT interval (QTc) >/= 470 msec.
* Clinically significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, congestive heart failure (new York Heart Association >Class 2), unstable angina, uncontrolled hypertension, or myocardial infarction within 6 months of Screening, or any Class 3 or 4 cardiac disease as defined by the New York Heart Association Functional Classification.
* Any uncontrolled active systemic infection or recent infection requiring intravenous anti-infective treatment that was complete ≤ 14 days before the first dose of study drug.
* Unresolved toxicities from prior anti-cancer therapy, defined as having not resolved to Common Terminology Criteria for Adverse Event (CTCAE, version 4.0), Grade 0 or 1, or to the levels dictated in the inclusion/exclusion criteria with the exception of alopecia.
* Known bleeding diathesis (e.g., von Willebrand's disease) or hemophilia.
* Known history of infection with human immunodeficiency virus (HIV) or history of active or chronic infection with hepatitis C virus (HCV) or hepatitis B virus (HBV), or any uncontrolled active systemic infection. Hepatitis B surface antigen must be confirmed negative within on year before enrollment. Subjects who are positive for hepatitis B core antibody or hepatitis B surface antigen must have a negative polymerase chain reaction (PCR) result before enrollment. Those who are PCR positive will be excluded.
* Any of the following abnormalities

  * Absolute neutrophil count (ANC) <750 cells/mm^3 (0.75 x 10^9/L)
  * Platelet count <50,000 cells/mm^3 (50 x 10^9/L) independent of transfusion support
  * Serum aspartate transaminase (AST) or alanine transaminase (ALT) ≥3.0 x upper limit of normal (ULN)
  * Creatinine clearance (CrCl) <30mL/min
  * Hemoglobin <8.0 g/dL
  * Bilirubin >1.5 x ULN (unless bilirubin rise is due to Gilbert's syndrome or of non-hepatic origin)
  * PT/INR >1.5 x ULN and PTT (aPTT) >1.5 x ULN(unless abnormalities are unrelated to coagulopathy or bleeding disorder).
* Unable to swallow capsules or disease significantly affecting gastrointestinal function such as malabsorption syndrome, resection of the stomach or small bowel, or complete bowel obstruction.
* Major surgery planned within 4 weeks of the first dose of study drug.
* Any life-threatening illness, medical condition, including uncontrolled diabetes mellitus (DM), or organ system dysfunction that, in the opinion of the investigator, could compromise the subject's safety or put the study outcomes at undue risk.
* Concurrent enrollment in another therapeutic investigational study or have previously taken ibrutinib.
* Lactating or pregnant.
* Unwilling or unable to participate in all required study evaluations and procedures.
* Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local subject privacy regulations).
* Currently active, clinically significant hepatic impairment Child-Pugh class B or C according to the Child Pugh classification.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2019-06-20 (Actual); Study Completion 2019-06-20 (Actual)

PRIMARY OUTCOMES:
Rate of conversion from FDG-PET positive to negative | 12 months
  The primary objective is to determine the rate of conversion from FDG-PET positive to negative at 12 months from the start of ibrutinib in patients receiving at least 6 months of Ibrutinib consolidation therapy for follicular lymphoma achieving at least a PR but remaining FDG-PET positive after first line chemoimmunotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Ariela Noy, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (9):
- United States (9):
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Center @ Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan - Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering at Mercy Medical Center, Rockville Centre, New York
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/